CLINICAL TRIAL: NCT03501446
Title: A Pilot Validation Study of Continuous CO2-based End-expiratory Lung Volume Measurements in Humans and an Experimental Porcine Model.
Brief Title: A Pilot Validation Study of Continuous CO2-based End-expiratory Lung Volume Measurements in Humans.
Acronym: ELVIS
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Tomas Öhman, Specialist in anaesthesia and intensive care, Karolinska Institutet
Other Study IDs: 2014/1393-31/2
Record Dates: First submitted 2018-04-10; First posted 2018-04-18 (Actual); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Ventilator Lung; Gas Exchange; Pulmonary Function
Keywords: PEEP optimization; Lung volumes

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The capnodynamic method non-invasively calculates effective lung volume (ELV) continuously during surgery. In this study ELV is compared to functionalresidual capacity (FRC) measured with Nitrogen Multiple Breath Wash out (NMBW) at 0 and 5 cm H2O Positive End Expiratory Pressure (PEEP) in patients scheduled for neck surgery at the Karolinska University Hospital, Solna, Sweden.

DETAILED DESCRIPTION:
The capnodynamic method continuously calculates effective lung volume (ELV) with the help of a capnodynamic equation:

ELV x (FACO2(n) - FACO2(n-1)) = delta t(n) x EPBF (CvCO2 - CvCO2(n)) - VTCO2. ELV Effective lung volume [L]. EPBF Effective pulmonary blood flow [L/min]. n current breath. n-1 previous breath. FACO2 mean alveolar carbon dioxide fraction. CvCO2 mixed venous carbon dioxide content [Lgas/Lblood]. CcCO2n pulmonary end-capillary carbon dioxide content [Lgas/Lblood]. VTCO2n volume [L] of carbon dioxide eliminated by the current, nth, breath. delta t n current breath cycle time [min]. The equation above describes the mole balance between the CO2 delivered to lungs (EPBF), the volume taking part in the gas exchange (ELV) and CO2 excreted from the lungs (VTCO2). Normally there is no difference in CO2 between the actual and the preceding breath as the same amount of CO2 as delivered to the lungs as is excreted. When small changes in CO2 concentration are inserted into the equation obtained with short inspiratory pauses in three out of nine breaths, nine different equations are obtained. The three unknown variables; ELV, EPBF and CvCO2 can be solved with a linear least square optimization, a well-known numerical mathematical principle. The breathing pattern is automatically controlled by the ventilator which provides continuous calculations of ELV where each value represents the average of the preceding nine breaths and renews with each breath as the newest replaces the oldest in the equation system.

At the day of surgery, included patients arrive at the surgical unit. After safe surgical checklist, vital signs are measured patients are anesthetized and muscle relaxed per routine practice. An endotracheal tube is inserted in the trachea and the patient connected to a ventilator. Anesthesia is maintained with Propofol in target controlled infusion and a short acting opioid is added as needed.

The protocol comprises a measurement of functional residual capacity (FRC) with the reference method, nitrogen multiple breath wash out (NMBW), at 0 cm H2O Positive End Expiratory Pressure (PEEP). The tracheal tube is then connected to the Servo-i ventilator with the capnodynamic breathing pattern applied. An ELV measurement at PEEP 0 cm H2O is followed by a measurement of ELV at PEEP 10 cm H2O and lastly a measurement of ELV at PEEP 5 cm H2O before the tube is clamped and connected to the NMBW reference method ventilator again for a measurement of FRC at PEEP 5 cm H2O.

The attending anesthesiologist has the final responsibility of the patient and could at any time end the protocol if needed.

ELIGIBILITY:
Inclusion Criteria:

* Individuals without current heart or lung disease

Exclusion Criteria:

* Obesitas
* Heart disease
* Lung disease
* Current smoker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals scheduled for neck surgery at Karolinska university hospital
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2014-12-01 (Actual); Primary Completion 2015-10-21 (Actual); Study Completion 2015-10-21 (Actual)

PRIMARY OUTCOMES:
Effective lung volume | Continous measurements during general anaesthesia and mechanical ventialtion, 45 minutes-2 hours
  Lung volume measurements during mechanical ventilation based on CO2 dynamics and a differentiated Fick's principle.

CONTACTS AND LOCATIONS:
Overall Officials: Håkan Björne, PhD, Study Director — Karolinska Institutet
Locations (1):
- Department of Perioperative Medicine and Intensive Care, Karolinska University Hospital, Solna, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided